CLINICAL TRIAL: NCT00095680
Title: A 24-week, Open-label Extension Study of the Efficacy, Safety, and Tolerability of Oral SCIO-469 in Treatment of Relapsed Refractory Patients With Multiple Myeloma
Brief Title: Extension Study of the Efficacy and Safety of Oral SCIO-469 in Relapsed, Refractory Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: VP Clinical Oncology, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005182; SCIO-469MMY2002 (B006)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; SCIO-469; Bortezomib; p38 MAP kinase
MeSH Terms: conditions — Multiple Myeloma | interventions — SCIO-469; Bortezomib

ARMS (2):
- 001 (Experimental): SCIO-469 two 30-mg capsules three times daily
  Interventions: Drug: SCIO-469
- 002 (Active Comparator): SCIO-469 and bortezomib The addition of bortezomib (treatment regimen or bolus) to monotherapy of SCIO-469 or bortezomib combination with SCIO-469 will be dependent upon clinical response or disease progression during the study
  Interventions: Drug: SCIO-469 and bortezomib

INTERVENTIONS:
Drug: SCIO-469 — two 30-mg capsules three times daily
  Arms: 001
Drug: SCIO-469 and bortezomib — The addition of bortezomib (treatment regimen or bolus) to monotherapy of SCIO-469 or bortezomib combination with SCIO-469 will be dependent upon clinical response or disease progression during the study
  Arms: 002

SUMMARY:
The main objective of this study is to assess the long-term effectiveness of SCIO-469 as monotherapy, or in combination with bortezomib in relapsed, refractory patients with multiple myeloma (MM) who have previously demonstrated clinical benefit in the Scios B003 study.

DETAILED DESCRIPTION:
The main objective of this study is to assess the long-term efficacy of SCIO-469 as monotherapy, or in combination with bortezomib in relapsed, refractory patients with multiple myeloma (MM) who have previously demonstrated clinical benefit in the Scios B003 study. Patients took by mouth two capsules (60 mg) three times a day alone or in combination with bortezomib, for 168 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not have disease progression on Day 73 of Study B003
* patients fully understand all elements of, and have signed and dated, the written Informed Consent Form (ICF) before initiation of protocol-specified procedures

Exclusion Criteria:

* Patients who have an active uncontrolled infection
* any condition, including laboratory abnormalities, that in the opinion of the investigator places the patient at unacceptable risk to participate in the study
* pregnant or lactating women, or who are not using adequate contraception
* sexually active women of childbearing potential (WCBP) who do not agree to use at least two forms of medically accepted birth control, including one barrier method, for the duration of the study
* men who do not agree to use an acceptable method for contraception throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Rate of response during therapy as measured by the European Group for Blood and Marrow Transplantation (EBMT) criteria. | Baseline to Day 168

SECONDARY OUTCOMES:
Time to first response and time to best response | Baseline, Wks 6,12,18,24, Day 198
Size and number of lytic bone lesions were summarized. | Baseline, Wks 6,12,18,24, Day 198
Pain was assessed by Pain Intensity Categorical Scale and Pain Intensity Visual Aid Scale. | Baseline, Wks 6,12,18,24, Day 198
Performance status was evaluated by Karnofsky scale. | Baseline, Wks 6,12,18,24, Day 198
Bone disease was monitored by assessing various biomarkers. | Baseline, Wks 6,12,18,24, Day 198
Number of patients with disease progression | Wks 6,12,18,24, Day 198

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.